CLINICAL TRIAL: NCT05220943
Title: The Effect of a Non-Operating Room Anesthesia (NORA) Safety Video on Clinician Anxiety and Perceived Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Louise Y. Wen, Principal Investigator, Staff Physician, Anesthesiology, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY02001332
Record Dates: First submitted 2022-01-06; First posted 2022-02-02 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Anxiety; Self Efficacy
MeSH Terms: conditions — Anxiety Disorders | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video (Other): All participants are invited to complete a pre survey, watch a five minute video, and then complete a post survey.
  Interventions: Behavioral: Video

INTERVENTIONS:
Behavioral: Video — This 5-minute video presents clips with voiceover narration summarizing and highlighting the key safety points in the Center for Surgical Innovation (CSI) location.

SUMMARY:
The purpose of this study is to assess the effect of a non-operating room anesthesia (NORA) safety video on clinician anxiety and perceived self-efficacy.

DETAILED DESCRIPTION:
50 anesthesia professionals will be recruited from the Center for Surgical Innovation (CSI) non-operating room anesthesia (NORA) workforce. Participants will be asked to: Complete a five-minute pre-survey, watch a five-minute video, and then complete a five-minute post-survey.

ELIGIBILITY:
Inclusion Criteria:

* Individuals employed at Dartmouth-Hitchcock Medical Center (DHMC) in the Department of Anesthesia who are eligible to work in the Center for Surgical Innovation (CSI).

Exclusion Criteria:

* Individuals who are not employed at Dartmouth-Hitchcock Medical Center (DHMC) in the Department of Anesthesia and who are not eligible to work in the Center for Surgical Innovation (CSI).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety | Before and after watching a five minute video, all occurring on the same day.
  Anxiety levels about working in the Center for Surgical Innovation (CSI) will be measured via a series of questions developed by the study team. The survey consist of multiple questions and responses include a scale; The options include "Not at all", "A little", "Moderately", "Very much" and "Extremely".

SECONDARY OUTCOMES:
Change in Perceived self-efficacy | Before and after watching a five minute video, all occurring on the same day.
  Perceived self-efficacy about working in the Center for Surgical Innovation (CSI) will be measured via a series of questions developed by the study team. The survey consist of multiple questions and responses include a scale; The options include "Not at all confident", "A little confident", "Moderately confident", "Very confident" and "Extremely confident".

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
There are not plans to make individual participant data available at this time.